CLINICAL TRIAL: NCT06403670
Title: The Effects of Dexmedetomidine and Remifentanil on Sedation and Comfort in Non-Operating Room Anesthesia: A Randomized, Double-blind, Controlled Trial
Brief Title: Dexmedetomidine and Remifentanil in NORA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University Ankara Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Uslu, MD, Research assistant, Baskent University Ankara Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NORADEX
Record Dates: First submitted 2024-05-01; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Comparison of the Effects of Remifentanil and Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Dex (Active Comparator): Group Dex received 0.5 mcg/kg of dexmedetomidine IV for 10 minutes, then dexmedetomidine infusion was started at 0.1-0.7 mcg/kg/h. Propofol 1 mg/kg was administered after waiting for 5 minutes for adequate sedation to develop due to dexmedetomidine's delayed onset of action.
  Interventions: Drug: Dexmedetomidine
- Group Remi (Active Comparator): Group RP received remifentanil 0.1 mcg/kg intravenously for 2 minutes, then remifentanil infusion was started at 0.01-0.1 mcg/kg/min. After waiting 2 minutes to develop a sufficient sedation level, 1 mg/kg of propofol was given.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Dexmedetomidine — Group DP received 0.5 mcg/kg of dexmedetomidine IV for 30 seconds, then dexmedetomidine infusion was started at 0.1-0.7 mcg/kg/h. Propofol 1 mg/kg was administered after waiting for 5 minutes for adequate sedation to develop due to dexmedetomidine's delayed onset of action.
  Arms: Group Dex
Drug: Remifentanil — Group RP received remifentanil 0.1 mcg/kg intravenously for 30 seconds, then remifentanil infusion was started at 0.01-0.1 mcg/kg/min. After waiting 2 minutes to develop a sufficient sedation level, 1 mg/kg of propofol was given.
  Arms: Group Remi

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) procedure is frequently encountered in non-operating room anesthesia applications (NORA). It is a procedure that requires deep sedation and analgesia in terms of gastroenterologist and patient comfort. Dexmedetomidine, which is increasingly used in NORA applications, comes to the fore because it does not cause respiratory depression, reduces the stress response, and provides hemodynamic stability. This study aims to compare the effects of dexmedetomidine-propofol (DP) and remifentanil-propofol (RP) combinations on hemodynamic stability, rapid recovery, and patient comfort in patients who underwent ERCP.

ELIGIBILITY:
Inclusion Criteria:

-ASA 1-3

Exclusion Criteria:

* Neurological disease,
* Psychiatric disease,
* Coronary artery disease,
* Long-term sedative drug use,
* Pregnant patients,
* Known allergy to planned drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-12-17 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Agitation-Sedation | 0 and 5 minutes after ERCP ends
  It will be evaluated with a Richmond Agitation-Sedation Scale.
Hemodynamic stability | 5, 10, 15, 25, 35. minutes
  Mean arterial pressure with non-invasive blood pressure monitoring (mmHg)

SECONDARY OUTCOMES:
Minimize drug dose | 5, 10, 15, 25, 35. minutes
  Amounts of medication administered throughout the procedure period will be collected.
Patient comfort | 30 minutes after ERCP ends
  It will be evaluated by nausea-vomiting and survey.
Rapid recovery | 30 minutes after ERCP ends
  It will be evaluated with a Modified Aldrete Score.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University Ankara Hospital, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No